CLINICAL TRIAL: NCT04442529
Title: Qatar Mothers and Babies: Examining the Feasibility, Acceptability, and Preliminary Outcomes Associated With Integrating a Postpartum Depression Intervention Into Perinatal Services for Women
Brief Title: Mothers and Babies Qatar (MB-Q): A Postpartum Depression Intervention
Acronym: MB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidra Medicine (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0004
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Postpartum Depression; Anxiety; Diabetes
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Pregnant women will receive prenatal care as usual.
- Intervention (Experimental): Pregnant women will receive the 12-session Mothers and Babies intervention
  Interventions: Behavioral: Mothers and Babies (MB)

INTERVENTIONS:
Behavioral: Mothers and Babies (MB) — Mothers and Babies is an evidence-based postpartum depression prevention intervention. It consists of 12 sessions which each last between 15-20 minutes. Intervention sessions are to be delivered either in person or by phone. The intervention is based on principles of cognitive-behavioral therapy (CBT).
  Arms: Intervention

SUMMARY:
Qatar Mothers and Babies is a 4-year collaboration between Northwestern University Feinberg School of Medicine and Sidra Medicine in Doha, Qatar that will generate and evaluate a cultural and contextual adaptation of the Mothers and Babies intervention for pregnant Arabic-speaking women in Qatar. The study will examine the feasibility and acceptability of the adapted intervention as well as its effectiveness in improving mental health outcomes among pregnant women receiving prenatal care at Sidra Medicine in Doha. Additionally, given the high prevalence of diabetes among this study population, the investigators are also interested in seeing if the Mothers and Babies interventions helps improve the management of this disease. Funded by the Qatar National Research Fund's National Priorities Research Program (NPRP), this project has the potential to guide future cultural adaptations of Mothers and Babies as well as other evidence-based interventions, and the delivery of Mothers and Babies to Arab and Arab-American women.

DETAILED DESCRIPTION:
Postpartum depression and anxiety are the two most common perinatal mental health disorders (mental health disorders occurring during pregnancy and the year after birth), with prevalence rates higher among women living in Qatar than in most western countries. The negative outcomes associated with postpartum depression and anxiety are profound, and include poor birth outcomes, poor parenting practices, and compromised infant and young child development. Although interventions exist to prevent postpartum depression and anxiety, to date there have been no studies that have attempted to prevent postpartum depression or anxiety among Arabic speaking women in the Middle East, including Qatar. This project brings together a multidisciplinary team of researchers and clinicians from Sidra Medicine (Qatar) and Northwestern University Feinberg School of Medicine (USA) to conduct a first-of-its-kind study that examines the feasibility, acceptability, and outcomes associated with an evidence-based postpartum depression intervention-Mothers and Babies (MB). MB has been widely used in the USA and has been linguistically translated into Arabic and successfully delivered to Arab-American women. In Phase One of this project, the investigators will culturally and contextually adapt Mothers and Babies to ensure its suitability for use with women residing in Qatar. In Phase Two, the investigators will conduct a small pilot study that examines the acceptability, appropriateness, and feasibility of the adapted Mothers and Babies intervention. Specifically, the investigators will deliver the adapted intervention to 10 women receiving prenatal care at Sidra Medicine. In Phase Three, the investigators will conduct a randomized controlled trial (n = 210) to determine the effectiveness of the adapted Mothers and Babies intervention on depressive symptoms, anxiety symptoms, and perceived stress among women receiving prenatal care at Sidra Medicine. As part of the randomized controlled trial, the investigators will recruit a sub-group of 40 women with diabetes, given the high prevalence of diabetes among women in Qatar and the negative outcomes associated with diabetes on mother and child. The investigators will explore whether the cognitive-behavioral techniques in Mothers and Babies are effective not only in promoting better mental health outcomes among this subgroup, but also better diabetes self-management.

ELIGIBILITY:
Inclusion criteria are identical for the pilot study and RCT.

* Participants must be 18 years of age or older
* Participants should speak Arabic fluently
* Participants must be up to 28 + 0 weeks pregnant
* Participants should not be diagnosed with a fetal anomaly that is incompatible with life or whose anomalies will have significant physical or developmental morbidity
* Participants should not be currently receiving treatment for mental health difficulties,
* Participants should not have a history of a serious mental health condition and,
* Participants must screen between 6-12 on the Edinburgh Postpartum Depression Scale (EPDS) and/or 5-14 on the Generalized Anxiety and Depression Scale (GAD-7).

Exclusion criteria:

* Participants who do not meet these screening criteria but are experiencing mild to moderate symptoms of depression will be provided mental health resources including a link to the Mothers & Babies website with English and Arabic manuals for self-directed study.
* Screened women scoring > 14 on the GAD-7 and/or >12 on the EPDS and/or those currently receiving mental health treatment will be offered a referral to Sidra's Women's Mental Health Clinic for further evaluation and treatment, as needed.
* Anyone who endorses the suicidality question ideation (EPDS #10) will be offered same day review by a Sidra women's mental health clinician, who will ascertain the level of risk and offer assistance as clinically indicated.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant female
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Pre-Screening tool
  First primary outcome of depressive symptoms is the Edinburgh Postpartum Depression Scale (EPDS). Scores are determined by participant self-report on screening questions. The total can range from 0 to 30 with higher scores indicating greater depressive symptoms.
Anxiety symptoms | Pre-Screening tool
  Second primary outcome of anxiety symptoms is the Generalized Anxiety Disorder 7-Item Scale (GAD-7). Scores are determined by participant self-report on screening questions. The GAD-7 total score can range from 0-21 with higher scores indicating more anxiety symptoms.
Perceived stress | Baseline and six month follow-up
  Third primary outcome of perceived stress is the Perceived Stress Scale 10-item version (PSS-10). Scores are determined by participant self-report at baseline and six-month follow-up. Scores range from 0-40 with higher scores indicate greater perceived stress.

SECONDARY OUTCOMES:
Behavioral Activation | Baseline and six month follow-up
  Behavioral Activation will be measured using the Behavioral Activation Depression Scale (BADS). The BADS assesses behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation strategies. It examines changes in the following areas: activation, avoidance/ rumination, work/school impairment, and social impairment. The BADS consists of 25 items, each rated on a seven point scale ranging from 0 (not at all) to 6 (completely). The range of the scale is 0-64. For the total scale, higher scores represent increased activation. The BADS has demonstrated strong internal consistency, construct validity, and predictive validity (Kanter et al, 2007; Kanter et al., 2009).
Mood Regulation | Baseline and six month follow-up
  Mood regulation will be measured using the 30-item Negative Mood Regulation Scale (NMRS) (Catanzaro & Means, 1990). For each question, participants will use a 5-point scale to indicate participants' beliefs, or when participants are disappointed or experiencing a negative mood. For the analyses, the study investigators will develop an average to these items to create a mean NMRS score (range 1-5). Higher scores indicate a greater ability to regulate one's mood.
Social Support | Baseline and six month follow-up
  Social support will be measured using the 19-item Medical Outcomes Study Social Support Survey (MOS-SSS) (Sherbourne & Stewart, 1991). This brief self-administered survey includes an overall functional social support index, as well as four functional support subscales: affectionate, emotional/informational, tangible, and positive social interaction. The range is 1-5 with greater scores indicating more perceived social support.
Decentering Thoughts | Baseline and six month follow-up
  Secondary outcome of Decentering will be measured using the Experiences Questionnaire (EQ) (Fresco et al., 2007). The EQ is a 20 item self-report scale designed to measure decentering and rumination, which has demonstrated strong internal consistency in a number of studies examining effects of interventions that incorporate cognitive restructuring techniques. Response choices are on a 1-5 scale. For the purposes of data analyses, study investigators will create a mean EQ score (range 1-5), with higher scores indicating more decentering/rumination.
Diabetes self-management | Baseline and six month follow-up
  The Diabetes self-care will be assessed using the summary of Diabetes Self-Management questionnaire. The tool contains 16 items, it is a reliable and valid instrument and enables an efficient assessment of self-care behaviors associated with glycemic control. Scale scores were calculated as sums of item scores and then transformed to a scale ranging from 0 to 10 (raw score / theoretical maximum score * 10). A transformed score of ten represents the highest self-rating of the assessed behavior.
Religious Coping- major life stressors | Baseline and six month follow-up
  The Religious Coping- major life stressors tool is a continuous scale which contains 12 items of religious coping with major life stressors. It has helped contributing to the growth of knowledge about the religion roles that serve in the process of dealing with crisis, trauma, and transition.
Mothers and Babies Skill Utilization | Six-month follow-up
  The Mothers and Babies Skill Utilization is administered at the 6-month follow-up survey with higher scores indicating greater use of in daily life. The instrument that will be utilized has been developed by the investigators.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidra, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
The investigators anticipate making the individual participant data available to other researchers who submit a reasonable request to analyze study data.

REFERENCES:
- [Derived] Ahmed SR, Watt F, Mahfoud ZR, Korayem M, Buhmaid S, Alberry M, Ibrahim IM, Tandon SD. Examining Feasibility, Acceptability, and Preliminary Outcomes of a Culturally Adapted Evidence-Based Postpartum Depression Preventive Intervention for Women in Doha, Qatar: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Aug 11;12:e11623. doi: 10.2196/11623. PMID 37566449